CLINICAL TRIAL: NCT07031726
Title: The Effectiveness of Worksite Nutrition and Wellness Program on Changes in Body Composition, Metabolic Profile, and Physical Fitness Among Employees
Brief Title: Effect of Nutrition and Wellness Program on Health Parameter Among Employees
Acronym: WNWP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Brawijaya (Other)
Collaborators: Universiti Putra Malaysia (Other); Universiti Teknologi MARA (UiTM) Sungai Buloh Campus, Malaysia (Unknown)
Responsible Party: Principal Investigator, Irka Dwi, Principal Investigator, University of Brawijaya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UBGizi2025WNWP01S2; UBStar Internal Grant (Other: Universitas Brawijaya - UBStar Program)
Record Dates: First submitted 2025-05-24; First posted 2025-06-22 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Obesity Prevention; Wellness Program; Body Composition; Nutrition; Workplace Interventions
Keywords: worksite wellness program; obesity prevention; personalized physical activity; personalized nutrition; employee health
MeSH Terms: interventions — Health Promotion

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to different groups based on faculty divisions using a cluster allocation model. Each group will receive either a structured wellness program or usual care.
Who Masked: Participant
Masking Description: Participants were blinded to group assignment to reduce bias in self-reported outcomes and compliance. Investigators and outcome assessors were not blinded due to the nature of the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Worksite nutrition and wellness program (Experimental): Participants receive a 12-week worksite nutrition and wellness program in a university setting. Core components include: (1) nutrition education sessions on healthy diet and portion control, (2) workplace-based wellness support and behavior-change strategies (e.g., goal setting and self-monitoring), and (3) physical activity component [e.g., brisk walking program/weekly targets]. Delivery mode: [group sessions/online messaging/face-to-face], frequency: [e.g., weekly/biweekly], and adherence support: [e.g., reminders, tracking, incentives if used]. Outcomes are assessed at baseline and post-intervention [plus interim assessments if applicable].
  Interventions: Behavioral: Worksite Nutrition and Wellness Program
- Standard Education Group (Active Comparator): Participants in this group will receive standard educational materials about nutrition and physical activity based on the official guidelines published by the Indonesian Ministry of Health. No structured or personalized intervention will be provided.
  Interventions: Behavioral: Standard education

INTERVENTIONS:
Behavioral: Worksite Nutrition and Wellness Program — A structured behavioral intervention combining personalized physical activity and structured physical activity (Zumba classes), personalized nutrition counseling, and mobile app-based self-monitoring.
  Other Names: WNWP; personalized physical activity; personalized nutrition
  Arms: Worksite nutrition and wellness program
Behavioral: Standard education — General educational materials on healthy eating and physical activity based on the Ministry of Health guidelines. No tailored or active intervention provided.
  Arms: Standard Education Group

SUMMARY:
This study aims to evaluate the effectiveness of a worksite-based nutrition and wellness program in improving body composition, metabolic profile, and physical fitness among university employees who are overweight or obese. The intervention includes personalized and structured physical activity (brisk walking), nutritional education, and self-monitoring using mobile applications. Participants will be assessed at baseline, after 6 weeks and 12 weeks of intervention to determine changes in fat mass, muscle mass, waist circumference, and related health indicators. This program is designed to promote healthier lifestyle habits and prevent non-communicable diseases in the workplace.

DETAILED DESCRIPTION:
This study is cluster randomized controlled trial conducted at Universitas Brawijaya to assess the effectiveness of a comprehensive workplace-based wellness intervention. The intervention comprises three key components: (1) structured physical activity is brisk walking with 150 minutes minimum for target per week; (2) personalized nutrition education delivered through interactive counseling; and (3) daily self-monitoring using a mobile application.

Participants include university employees categorized as overweight or obese, who work in sedentary office jobs for more than 5 hours per day. Subjects will be assessed at three time points-baseline, after 6 weeks, and after 12 weeks-to measure changes in body composition (e.g., body mass index, body fat percentage, subcutaneous fat, skeletal mass, and waist circumference), metabolic profile (e.g., fasting blood glucose and cholesterol), and physical fitness parameters.

The study aims to provide evidence on the impact of structured, low-cost wellness programs in reducing obesity-related health risks among adult employees in institutional settings. Ethical approval has been obtained from the Faculty of health, Universitas Brawijaya. The results are expected to support future implementation of health promotion policies in the workplace.

ELIGIBILITY:
Inclusion Criteria:

* Employees aged 20-40 years
* BMI ≥ 23 kg/m²
* Body fat percentage ≥ 25% as measured by body composition analysis
* Employed in white-collar occupations with predominantly sedentary work activities, defined as sitting for ≥ 5 hours per day, based on results from the Global Physical Activity Questionnaire (GPAQ).
* Not engaging in regular vigorous physical activity, defined as participating in such activity less than 3 times per week, according to GPAQ results.
* Not having a medical condition that could inhibit participation in the intervention.
* Be willing to attend the program for a full 12 weeks.

Exclusion Criteria:

* A history of severe chronic disease, including type 1 diabetes, severe coronary heart disease, or kidney failure.
* Be enrolled in other weight loss programs that may affect the results of the study.
* Regular engagement in vigorous-intensity exercise prior to the start of the intervention program.
* Not classified as a white-collar sedentary worker based on the Global Physical Activity Questionnaire (GPAQ) assessment.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 98 (Actual)
Dates: Start 2025-06-12 (Actual); Primary Completion 2025-10-02 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Change in Body Mass Index (BMI) | Baseline, Week 6, and Week 12
  Change in BMI measured using standard anthropometric protocol

SECONDARY OUTCOMES:
Body Fat Percentage | At Baseline, Week 6, and Week 12
  % Body fat in percentage measured via bioelectrical impedance analysis (BIA).
Skeletal mass | Baseline, week 6, Week 12
  Skeletal mass in percentage using BIA.
Change in Waist Circumference | Baseline, Week 6, Week 12
  Waist measured in centimeters at midpoint between lowest rib and iliac crest.
Change in Hand Grip Strength | Baseline, Week 6, and Week 12
  Measured using a digital dynamometer (dominant hand).
Change in VO₂ Max | Baseline, Week 6, and Week 12
  Estimated VO₂ Max via submaximal aerobic capacity test (e.g., Rockport or Queens step test).
Change in Fasting Blood Glucose | Baseline and Week 12
  Measured using capillary blood sample with a point-of-care glucometer (EasyTouch®) after ≥8 hours fasting.
Change in Total Blood Cholesterol | Baseline and Week 12
  Total cholesterol measured using capillary blood with a point-of-care cholesterol meter (EasyTouch®).

CONTACTS AND LOCATIONS:
Overall Officials: Irka Dwi Fatmawati, S.Tr. Gz., Principal Investigator — University of Brawijaya
Locations (1):
- Universitas Brawijaya - Kampus 2, Malang, East Java, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD), including anthropometric measurements (BMI, body composition, waist circumference), hand grip strength, VO₂ max estimates, and fasting glucose and cholesterol levels will be shared.
Supporting Information: Study Protocol, ICF
Time Frame: The data will be available beginning 6 months after study completion and will remain accessible for up to 3 years.
Access Criteria: Access will be granted to qualified researchers upon reasonable request. The data will be shared in de-identified format via secure email or institutional data repository, pending ethical approval and data use agreement.